CLINICAL TRIAL: NCT00069264
Title: A Phase I Dose-Finding Study of E7389 (Halichondrin B Analog) in Patients With Advanced Solid Tumors
Brief Title: Study of E7389 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-101; E7389; BOLD
Record Dates: First submitted 2003-09-19; First posted 2003-09-24 (Estimated); Results first posted 2011-12-20 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-11

CONDITIONS: Advanced Solid Tumors
Keywords: Metastatic Tumors; Advanced Solid Tumors; Stage IV Tumors; Solid Tumors; Recurrent Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — eribulin

ARMS (1):
- E7389 (Experimental)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — E7389 Dose-escalation starting at 0.25 mg/m^2 intravenous on Days 1, 8, and 15 of a 28 day cycle.

SUMMARY:
To determine the maximum tolerated dose of E7389 in patients with advanced solid tumors that have progressed following standard therapy or for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a histologically or cytologically confirmed and measurable advanced solid tumor that has progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy)
* Patients may have received prior chemotherapy
* Patients must be aged > 18 years
* Patients must have a Karnofsky Performance Status of > 70%
* Patients must have a life expectancy of > 3 months
* Patients must have adequate renal function as evidenced by serum creatinine <1.5mg/dL or creatinine clearance >= 45mL/minute
* Patients must have adequate bone marrow function as evidenced by absolute neutrophil count > 1,500/µL and platelets > 100,000/µL
* Patients must have adequate liver function as evidenced by bilirubin < 1.5mg/dL and alanine transaminase (ALAT) and aspartate transaminase (ASAT) <= 2 times the upper limits of normal (ULN)unless related to liver involvement by tumor, in which case <= 5.0 times ULN
* Patients must be willing and able to comply with the study protocol for the duration of the study
* Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice

Exclusion Criteria

* Patients who have received chemotherapy within three weeks (six weeks if nitrosoureas were received) of E7389 treatment start
* Patients who have not recovered from any chemotherapy related or other therapy related toxicity at study entry
* Patients who require active anti-coagulant therapy
* Women who are pregnant or breastfeeding. Women of childbearing potential with either a positive pregnancy test at Screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential)
* Fertile men who are not willing to use contraception or fertile men with a female partner who is not willing to use contraception
* Patients who have not successfully completed local therapy for previously treated central nervous system (CNS) metastases and who have not been discontinued from corticosteroids for at least four weeks before starting treatment with E7389. Patients with asymptomatic brain metastases who have no evidence of midline shift on CT scan or MRI may be enrolled without initiation of local therapy for the CNS metastases. In this case, a repeat scan must be performed within four weeks of the original scan to ensure that disease progression is not occurring.
* Patients who have tested positive for HIV
* Patients with severe uncontrolled intercurrent illness/infection (excluding malignancies)
* Patients with uncontrolled cardiovascular illness defined as unstable angina, myocardial infarction within 6 months prior to study entry, symptomatic congestive heart failure (CHF) (NYHA II or higher) clinical evidence of CHF, or clinical evidence of serious cardiac arrhythmia
* Patients with organ allografts
* Patients who have received investigational drugs, including immunotherapy, gene therapy, hormone therapy, or other biologic therapy; anti-neoplastic therapy; or radiation therapy (other than required for palliation) within three weeks of E7389 treatment start
* Patients who have had major surgery within four weeks of E7389 treatment start without a full recovery
* Patients with a hypersensitivity to Halichondrin B and/or Halichondrin B-like compounds
* Patients with other significant disease that, in the Investigator's opinion, would exclude the patient from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-09; Primary Completion 2005-03 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Shuster, Ph.D., Study Director — Eisai Inc.
Locations (2):
- United States (2):
  - The Bronx, New York
  - San Antonio, Texas

REFERENCES:
- See also: Related Info — http://www.eisai.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E7389
Started | 32
Completed | 0
Not Completed | 32
Not completed — Adverse Event | 3
Not completed — Progressive Disease | 23
Not completed — Withdrawal by Subject | 3
Not completed — Discon Therapy | 3

BASELINE CHARACTERISTICS:
Arm/Group | E7389
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Please note: 8 subjects in unknown category were Hispanic/Latino
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 7
    White | 16
    More than one race | 0
    Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose
Time Frame: 28 Days
Measure: Number; unit: mg/m^2
Arm/Group | E7389
Number analyzed (Participants) | 32
mg/m^2 | 1.0

ADVERSE EVENTS:
Arm/Group | E7389
Serious Adverse Events (participants affected / at risk) | 12/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 (N=32)
Ascites (Gastrointestinal disorders) | 3
Chest Pain (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Klebsiella Infection (Infections and infestations) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Pain (General disorders) | 1
Fatigue (General disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Anoxic Encephalopathy (Nervous system disorders) | 1
Multi-Organ System Failure (General disorders) | 1
Sepsis (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Catheter Related Infection (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 (N=32)
Anemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 9
Palpitations (Cardiac disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 14
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 8
Chest Pain (General disorders) | 2
Fatigue (General disorders) | 19
Peripheral Edema (General disorders) | 4
Pain (General disorders) | 2
Pyrexia (General disorders) | 5
Aspartate Aminotransferase Increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Neuropathy (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No